CLINICAL TRIAL: NCT00689000
Title: A Phase I-II Study to Evaluate the Safety, Tolerability and Anti-Disease Activity of the Aminopeptidase Inhibitor, CHR-2797, in Elderly and/or Treatment Refractory Patients With Acute Myeloid Leukemia or Multiple Myeloma
Brief Title: Safety and Anti-Disease Activity of CHR-2797 (Tosedostat) in Elderly and/or Treatment Refractory Patients With Acute Myeloid Leukemia (AML) and Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Dr Leon Hooftman, Chief Medical Officer, Chroma Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2797-002
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: Leukemia; AML; MDS; MM; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Multiple Myeloma; Cancer; Hematological malignancies; Elderly; Refractory; Blood
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Multiple Myeloma; Leukemia; Neoplasms; Hematologic Neoplasms | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CHR-2797 (tosedostat) (Experimental): oral, once daily administration of CHR-2797 to determine safety & anti-disease activity.
  Interventions: Drug: CHR-2797 (tosedostat): Aminopeptidase inhibitor

INTERVENTIONS:
Drug: CHR-2797 (tosedostat): Aminopeptidase inhibitor — Phase I: Once daily, oral ingestion of CHR-2797 capsules (60mg, 90mg, 130mg or 180mg) depending on cohort
  Phase II: Once daily, oral ingestion of 130mg CHR-2797 (recommended dose from Phase I) until progressive disease or withdrawal from the study
  Other Names: tosedostat; CHR-2797; aminopeptidase inhibitor

SUMMARY:
This is an open-label, non-randomised, multi-centre phase I-II study of CHR-2797 administered orally once a day. The study involves two distinct phases:

* Phase I: an open-label, dose-escalating phase of the study to explore the safety, tolerability, and pharmacokinetics (PK) of CHR-2797.
* Phase II: the recommended dose level of CHR-2797, as determined in phase I, will be administered to a further cohort of approximately 40 patients to determine whether CHR-2797 has sufficient biological activity against the disease(s) under study.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, multi-centre phase I-II study of CHR-2797 administered orally once a day. The study involves two distinct phases:

Phase I: an open-label, dose-escalating phase of the study to explore the safety, tolerability, and pharmacokinetics (PK) of CHR-2797. Cohorts of 3-6 patients each will be treated with escalating, once daily, oral doses of CHR-2797 for 84 days (12 weeks), of which the first 28 days constitute the dose finding/ DLT phase. The starting dose will be 60 mg once daily. Doses will be increased in a stepwise fashion by around 40 percent per step until the MTD is reached. The proportion of patients with Multiple Myeloma will be limited to one third: one per cohort of 3 or 2 per cohort of 6. It is anticipated that 24-30 patients will be enrolled in the phase I portion of the trial. A decision will be made with regard to the disease indication to be tested in phase II (either AML/MDS or MM or both), after completion of phase I, or following definition of MTD.

Phase II: the recommended dose as determined in phase I, will be administered for 84 days to a maximum of 40 patients. The primary objective is to determine whether CHR-2797 has sufficient biological activity against the disease(s) under study. A multinomial stopping rule has been included in the design that incorporates objective responses and early progression into a decision to stop or continue this phase I/II trial. An interim assessment will be performed after 15 patients have received the maximum acceptable dose (MAD) dose of CHR-2797 with clearly defined early stopping rules.

There will be a clinical conference at the end of every cohort in the phase I portion of the study, between phase I and II and after the first 15 patients have completed therapy in phase II.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent.
* Patients with AML, MDS (subtype RAEB-1 or RAEB-2), or MM whose disease has relapsed or is refractory to front line and/ or salvage therapy; elderly patients (≥ 60 years) with AML, MDS, MM who are not candidates for chemotherapy and for whom other therapy is inappropriate.
* Patients should have recovered from the acute adverse effects of prior therapies (excluding alopecia and grade II neuropathy).
* AML, MDS and MM are diseases of the haematopoietic system and can cause myelosuppression. Consequently supportive therapy should be given to ensure adequate values, according to local guidelines.
* A bone marrow aspirate/ biopsy performed within four weeks prior to study entry.
* Adequate bone marrow, hepatic and renal function including the following:

  1. Patients with high blast counts can be included in the trial, if they can be controlled by the use of hydroxyurea (500-3000 mg daily).
  2. Total bilirubin ≤ 1.5 x upper normal limit.
  3. AST (SGOT), ALT (SGPT) ≤ 2.5 x upper normal limit.
  4. Creatinine ≤1.5 x upper normal limit.
* Age ≥ 18 years
* Performance status (PS) ≤ 2 (ECOG scale).
* Estimated life-expectancy greater than 3 months.
* Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of the trial. A woman with reproductive potential is defined as one who is biologically capable of becoming pregnant. Patients who are not surgically sterile or postmenopausal must agree to use a medically acceptable and highly effective method of birth control for the duration of the study and to continue after the end of CHR-2797 treatment for a further 3 months (female patients) or for a further 6 months (for male patients and their partners). A highly effective method of birth control is defined as any method that results in a low failure rate, including implants, injectables, some intra-uterine devices (IUD's), sexual abstinence, and vasectomy/ sterilization. Sexually active males and females using oral contraceptive pills should also use barrier contraception. Although there is no reason to believe that the use of CHR-2797 has an effect on the pharmacokinetics of hormonal contraceptives, this has not yet been proven.

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to trial entry- except for hydroxyurea (maximum daily dose is 3 g).
* Indolent, smouldering myeloma, monoclonal gammopathy with unknown significance.
* Patients who need a daily dose of hydroxyurea greater than 3 g to control leukocytosis.
* Co-existing active infection or serious concurrent illness.
* Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.
* Gastrointestinal disorders that may interfere with absorption of the study drug.
* Patients with platelet count(s) < 20,000.
* Patients who have had a blood transfusion (platelet support or packed cells) within 7 days prior to study entry.
* Persistent grade II or greater toxicity from any cause (except haematological toxicities and peripheral neuropathy).
* Patients with grade III-IV peripheral neuropathy.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Phase I: To determine the safety, tolerability, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of CHR-2797 when administered orally, once daily. | first 28 days of treatment
Phase II: To evaluate the anti-leukaemia/myeloma effect of the recommended dose of single agent CHR-2797. | End of study

SECONDARY OUTCOMES:
Phase I and II: To determine trough levels of CHR-2797 when administered orally, once daily, at different dose levels. | End of study
Phase II: To evaluate the safety and tolerability of the recommended dose of CHR-2797 when administered orally, once daily. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Morgan, MD, Principal Investigator — Royal Marsden Hospital, UK; Gert Ossenkoppele, MD, Principal Investigator — Vrije Universiteit MC, Amsterdam; Pierre Zachée, MD, Principal Investigator — ZNA Antwerpen, Belgium; Alan Burnett, MD, Principal Investigator — University Hospital, Cardiff, United Kingdom; Michel Delforge, MD, Principal Investigator — UZ Gasthuisberg, Leuven, Belgium; Bob Lowenberg, MD, Principal Investigator — Erasmus MC, Rotterdam; Ulrich Dührsen, MD, Principal Investigator — Universitätsklinikum, Essen, Germany; Carsten Müller-Tidow, MD, Principal Investigator — Universitätsklinikum, Münster, Germany
Locations (1):
- Nexus Oncology Ltd, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Lowenberg B, Morgan G, Ossenkoppele GJ, Burnett AK, Zachee P, Duhrsen U, Dierickx D, Muller-Tidow C, Sonneveld P, Krug U, Bone E, Flores N, Richardson AF, Hooftman L, Jenkins C, Zweegman S, Davies F. Phase I/II clinical study of Tosedostat, an inhibitor of aminopeptidases, in patients with acute myeloid leukemia and myelodysplasia. J Clin Oncol. 2010 Oct 1;28(28):4333-8. doi: 10.1200/JCO.2009.27.6295. Epub 2010 Aug 23. PMID 20733120